CLINICAL TRIAL: NCT02747875
Title: The Effect of Methadone vs. Fentanyl Administration on Postoperative Pain Control in Pediatric Patients Undergoing Cardiac Surgery: A Randomized, Double-Blinded Controlled Trial
Brief Title: Methadone vs. Fentanyl Administration on Postoperative Pain Control in Pediatric Patients Undergoing Cardiac Surgery
Acronym: CV_RCT_M_F
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Drug Shortage
Sponsor: Andrew Waberski (Other)
Responsible Party: Sponsor-Investigator, Andrew Waberski, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7364
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Opioid Use, Unspecified
Keywords: pediatric; cardiac bypass surgery; methadone; fentanyl; morphine
MeSH Terms: interventions — Methadone; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control - Fentanyl (Active Comparator): Participants will receive 20 mcg/kg of fentanyl prior to surgical incision, over 20 minutes. The medication will be prepared as described and all research and staff personnel as well as the study participant will be blinded to treatment group assignment.
  Interventions: Drug: Fentanyl
- Treatment - Methadone (Active Comparator): Participants will receive 0.3 mg/kg of methadone prior to surgical incision, over 20 minutes. The medication will be prepared as described and all research and staff personnel as well as the study participant will be blinded to treatment group assignment.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — The treatment phase will begin at the induction of general anesthesia and finish at the end of the surgical procedure. Under the direction of the cardiac anesthesiologist subjects will be premedicated and general anesthesia will be induced with standard anesthetic monitoring and management. Participants will receive 0.3 mg/kg of methadone prior to surgical incision, over 20 minutes. General anesthesia will be maintained with inhalational anesthetics and paralytics. The subject will continue to be evaluated for hemodynamic stability, bleeding, and respiratory effort. The postoperative intensive care phase will begin at time of room admission and end at day three of hospital stay. All subjects will receive morphine or oxycodone analgesics and sedation medication based on the hospital's postoperative pain control and agitation protocol. Standard electronic documentation will be maintained throughout and include: medications, vital signs, and events.
  Arms: Treatment - Methadone
Drug: Fentanyl — The treatment phase will begin at the induction of general anesthesia and finish at the end of the surgical procedure. Under the direction of the cardiac anesthesiologist subjects will be premedicated and general anesthesia will be induced with standard anesthetic monitoring and management. Participants will receive 20 mcg/kg of fentanyl prior to surgical incision, over 20 minutes. General anesthesia will be maintained with inhalational anesthetics and paralytics. The subject will continue to be evaluated for hemodynamic stability, bleeding, and respiratory effort. The postoperative intensive care phase will begin at time of room admission and end at day three of hospital stay. All subjects will receive morphine or oxycodone analgesics and sedation medication based on the hospital's postoperative pain control and agitation protocol. Standard electronic documentation will be maintained throughout and include: medications, vital signs, and events.
  Other Names: Sublimaze
  Arms: Control - Fentanyl

SUMMARY:
The purpose of this study is to determine if methadone improves postoperative pain control in pediatric patient's undergoing cardiac surgery.

DETAILED DESCRIPTION:
The proposed study will be conducted at Children's National Health System (CNHS). Pediatric subjects undergoing cardiac surgery requiring cardiopulmonary bypass will be recruited. Eligible and consenting participants will be assigned a unique identification number and will be randomly assigned to receive either methadone or fentanyl using a computer-generated randomization scheme. A total of 52 participants will be enrolled to each arm of the study, providing 80% power to detect a 30% difference between groups.

Once informed consent is obtained the inpatient pharmacist at CNHS will randomly assign eligible participants to receive methadone or fentanyl. The pharmacist will prepare 0.3 mcg/kg of methadone and 20 mcg/kg of fentanyl for loading dose administration, diluted to 10 mL.

The IDS pharmacy will store and maintain all medications per Department of Pharmacy standard operating procedures for waste of a controlled substance (C-II) drug.

The treatment phase will begin at the induction of general anesthesia and finish at the end of the surgical procedure. Standard anesthetic practice for monitoring, induction, and maintenance of general anesthesia will be preserved throughout.

Participants will receive either 0.3 mg/kg of methadone or 20 mcg/kg of fentanyl prior to surgical incision, over 20 minutes. The medication will be prepared as described above and all research and staff personnel as well as the study participant will be blinded to treatment group assignment.

As per standard anesthetic practice, the subject will continue to be evaluated for hemodynamic stability, postoperative risk of bleeding, and respiratory effort. Morphine at 0.05 mg/kg per dose will be administered intravenously as needed for pain control. Surgical procedures and times will be recorded in the operative report via the electronic medical record.

Postoperative ICU Phase The postoperative cardiac intensive care unit phase will begin at admission to the Cardiac Intensive Care Unit (CICU) and will end on the third day of hospital admission. Postoperative care including hemodynamic stability, resuscitation, and respiratory support will be at the discretion of the CICU team.

As per CICU protocol, the nurse will monitor and record vital signs and pain scale (FLACC) scores beginning at handoff from the anesthesia team to the intensive care team. The nurse will continue to document vital signs including: blood pressure, heart rate, respiratory rate, oxygen saturation, temperature, minute ventilation when mechanically ventilated, and oxygen supplementation when appropriate, in the electronic medical record every hour. As per nursing protocol, FLACC scores will be recorded in the electronic medical record every 4 hours or when the nursing staff witnesses pain during the entirety of the subject's CICU stay.

All subjects will receive analgesics and sedation medication based on CICU postoperative pain control and agitation protocol

Data Collection The investigator or designee, blinded to group assignment, will collect all of the relevant data from the electronic medical record within six months of the cardiac surgery and enter it into the Medical Center's proprietary web-based data-entry and data-management system, REDcap (Research Electronic Data Capture). The source of information will be medical records at the Children's National Health System "Anesthesiology" and "Bear Tracks" information systems provided by Cerner Corporation.

Data will be obtained specifically for research purposes. Subject identifiers (e.g. name, date of birth, address) will not be entered into the REDcap system. The previously assigned unique identification numbers will be used.

Statistical Considerations Significance will be measured as a 30% reduction in postoperative pain requirement. Statistical analysis will be used to evaluate any differences between the randomization groups in opioid-related adverse events during the first 24-hour postoperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 2 years and less than 8 years at the time of randomization.
2. Weight greater than 6 kg.
3. American Society of Anesthesiologists (ASA) physical status of ASA I, II, or III (Appendix I).
4. Informed consent to participate from the parent or legally authorized guardian.
5. Scheduled for congenital cardiac bypass surgery.

Exclusion Criteria

Subjects will not be eligible to participate in the study if any of the following exclusion criteria apply:

1. History or a family (parent or sibling) history of malignant hyperthermia.
2. Known significant hepatic disorders determined by medical history, medical record documentation, physical examination, or laboratory tests obtained during the routine preoperative cardiac surgery evaluation or cardiology visit (International Normalized Ratio (INR)>1.5).
3. Emergency Cardiac Surgery.
4. History of chronic nausea and/or vomiting.
5. Currently receiving inotropic agents or using a pacemaker.
6. Prexisting long QTc interval of greater than 460ms determined by medical history, medical record documentation, or electrocardiogram obtained during the routine preoperative cardiac surgery evaluation.
7. History of documented pulmonary hypertension, respiratory dysfunction, or requirement of supplemental oxygen therapy.
8. History of opioid abuse, addiction, or tolerance.
9. Obesity defined as a body weight greater than 130% of the ideal weight.
10. Participation in another clinical trial or any study that may interfere with participation in this trial.
11. History of allergic reaction to methadone or fentanyl.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Waberski, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barletta JF. Clinical and economic burden of opioid use for postsurgical pain: focus on ventilatory impairment and ileus. Pharmacotherapy. 2012 Sep;32(9 Suppl):12S-8S. doi: 10.1002/j.1875-9114.2012.01178.x. PMID 22956490
- [Result] Oderda G. Challenges in the management of acute postsurgical pain. Pharmacotherapy. 2012 Sep;32(9 Suppl):6S-11S. doi: 10.1002/j.1875-9114.2012.01177.x. PMID 22956493
- [Result] Lee LA, Caplan RA, Stephens LS, Posner KL, Terman GW, Voepel-Lewis T, Domino KB. Postoperative opioid-induced respiratory depression: a closed claims analysis. Anesthesiology. 2015 Mar;122(3):659-65. doi: 10.1097/ALN.0000000000000564. PMID 25536092
- [Result] Chia YY, Liu K, Wang JJ, Kuo MC, Ho ST. Intraoperative high dose fentanyl induces postoperative fentanyl tolerance. Can J Anaesth. 1999 Sep;46(9):872-7. doi: 10.1007/BF03012978. PMID 10490157
- [Result] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Result] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Result] Naguib AN, Tobias JD, Hall MW, Cismowski MJ, Miao Y, Barry N, Preston T, Galantowicz M, Hoffman TM. The role of different anesthetic techniques in altering the stress response during cardiac surgery in children: a prospective, double-blinded, and randomized study. Pediatr Crit Care Med. 2013 Jun;14(5):481-90. doi: 10.1097/PCC.0b013e31828a742c. PMID 23644384
- [Result] Bowdle TA, Even A, Shen DD, Swardstrom M. Methadone for the induction of anesthesia: plasma histamine concentration, arterial blood pressure, and heart rate. Anesth Analg. 2004 Jun;98(6):1692-1697. doi: 10.1213/01.ANE.0000114085.20751.20. PMID 15155330
- [Result] Ward RM, Drover DR, Hammer GB, Stemland CJ, Kern S, Tristani-Firouzi M, Lugo RA, Satterfield K, Anderson BJ. The pharmacokinetics of methadone and its metabolites in neonates, infants, and children. Paediatr Anaesth. 2014 Jun;24(6):591-601. doi: 10.1111/pan.12385. Epub 2014 Mar 26. PMID 24666686
- [Result] Udelsmann A, Maciel FG, Servian DC, Reis E, de Azevedo TM, Melo Mde S. Methadone and morphine during anesthesia induction for cardiac surgery. Repercussion in postoperative analgesia and prevalence of nausea and vomiting. Rev Bras Anestesiol. 2011 Nov-Dec;61(6):695-701. doi: 10.1016/S0034-7094(11)70078-2. English, Multiple languages. PMID 22063370
- [Result] Lee M, Silverman SM, Hansen H, Patel VB, Manchikanti L. A comprehensive review of opioid-induced hyperalgesia. Pain Physician. 2011 Mar-Apr;14(2):145-61. PMID 21412369
- [Result] Davis AM, Inturrisi CE. d-Methadone blocks morphine tolerance and N-methyl-D-aspartate-induced hyperalgesia. J Pharmacol Exp Ther. 1999 May;289(2):1048-53. PMID 10215686
- [Result] Liu JG, Liao XP, Gong ZH, Qin BY. The difference between methadone and morphine in regulation of delta-opioid receptors underlies the antagonistic effect of methadone on morphine-mediated cellular actions. Eur J Pharmacol. 1999 Jun 4;373(2-3):233-9. doi: 10.1016/s0014-2999(99)00270-8. PMID 10414444
- [Result] Bastero P, DiNardo JA, Pratap JN, Schwartz JM, Sivarajan VB. Early Perioperative Management After Pediatric Cardiac Surgery: Review at PCICS 2014. World J Pediatr Congenit Heart Surg. 2015 Oct;6(4):565-74. doi: 10.1177/2150135115601830. PMID 26467871
- [Result] Lotsch J. Pharmacokinetic-pharmacodynamic modeling of opioids. J Pain Symptom Manage. 2005 May;29(5 Suppl):S90-103. doi: 10.1016/j.jpainsymman.2005.01.012. PMID 15907650
- [Result] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Marymont JH, Shear T, Parikh KN, Patel SS, Gupta DK. Intraoperative Methadone for the Prevention of Postoperative Pain: A Randomized, Double-blinded Clinical Trial in Cardiac Surgical Patients. Anesthesiology. 2015 May;122(5):1112-22. doi: 10.1097/ALN.0000000000000633. PMID 25837528
- [Result] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Result] Gourlay GK, Willis RJ, Lamberty J. A double-blind comparison of the efficacy of methadone and morphine in postoperative pain control. Anesthesiology. 1986 Mar;64(3):322-7. doi: 10.1097/00000542-198603000-00004. PMID 3954126
- [Result] Gourlay GK, Willis RJ, Wilson PR. Postoperative pain control with methadone: influence of supplementary methadone doses and blood concentration--response relationships. Anesthesiology. 1984 Jul;61(1):19-26. PMID 6742480
- [Result] Berde CB, Beyer JE, Bournaki MC, Levin CR, Sethna NF. Comparison of morphine and methadone for prevention of postoperative pain in 3- to 7-year-old children. J Pediatr. 1991 Jul;119(1 Pt 1):136-41. doi: 10.1016/s0022-3476(05)81054-6. PMID 2066846
- [Result] Stemland CJ, Witte J, Colquhoun DA, Durieux ME, Langman LJ, Balireddy R, Thammishetti S, Abel MF, Anderson BJ. The pharmacokinetics of methadone in adolescents undergoing posterior spinal fusion. Paediatr Anaesth. 2013 Jan;23(1):51-7. doi: 10.1111/pan.12021. Epub 2012 Sep 14. PMID 22978825
- [Result] Voepel-Lewis T, Zanotti J, Dammeyer JA, Merkel S. Reliability and validity of the face, legs, activity, cry, consolability behavioral tool in assessing acute pain in critically ill patients. Am J Crit Care. 2010 Jan;19(1):55-61; quiz 62. doi: 10.4037/ajcc2010624. PMID 20045849
- [Result] Moss AJ. Measurement of the QT interval and the risk associated with QTc interval prolongation: a review. Am J Cardiol. 1993 Aug 26;72(6):23B-25B. doi: 10.1016/0002-9149(93)90036-c. PMID 8256751
- [Result] Price LC, Wobeter B, Delate T, Kurz D, Shanahan R. Methadone for pain and the risk of adverse cardiac outcomes. J Pain Symptom Manage. 2014 Sep;48(3):333-42.e1. doi: 10.1016/j.jpainsymman.2013.09.021. Epub 2014 Jan 28. PMID 24480532
- Available data/document: Study Protocol: Pr 7364 — http://www.irbear.org — The Effect of Methadone vs. Fentanyl Administration on Postoperative Pain Control in Pediatric Patients Undergoing Cardiac Surgery. A Randomized, Double-Blinded Controlled Trial

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was terminated because enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. Additionally, without notice formulations of the study drug methadone became unavailable and remain unavailable due to production shortages.
Period: Overall Study
Arm/Group | Control - Fentanyl | Treatment - Methadone
Started | 12 | 14
Completed | 11 | 13
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Fentanyl | Treatment - Methadone | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 14 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 4.1 [0.3 to 7.1] | 4.4 [2.3 to 7.8] | 4.2 [0.3 to 7.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 14 | 26

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Dose, in Morphine Equivalents, in the First 24 Hours After Pediatric Cardiac Bypass Surgery.
Description: The distribution of the total opioid dose in the first 24 hours will be evaluated by randomization group (methadone vs. fentanyl) and differences between groups will be tested. It is hypothesized that compared to fentanyl, methadone administered intraoperative will result in a significantly lower total opioid dose (morphine or oxycodone) during the first 24 hour postoperative period. Assuming no difference between the two treatment strategies in the population, a total sample size of 52 in each group will provide 80% power to detect an effect size of 0.1. Significance will be measured as a 30% reduction in postoperative pain requirement.
Time Frame: 24 hours
Population: The trail was terminated because enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. Additionally, without notice formulations of the study drug methadone became unavailable and remain unavailable due to production shortages. Therefore, no analysis was performed on the data.
Measure: Mean (Standard Deviation); unit: mg postop morphine equivelant 24hr
Arm/Group | Control - Fentanyl | Treatment - Methadone
Number analyzed (Participants) | 11 | 13
mg postop morphine equivelant 24hr | 0.55 (0.21) | 0.48 (0.24)

2. Secondary Outcome: Opioid-related Adverse Events Including: Respiratory Failure, Cardiovascular Instability, and Postoperative Nausea and Vomiting
Description: Opioid-related adverse events will be monitored closely and a secondary analysis will compare the incidence of side effects between the two groups during the first 24-hour postoperative period. The Pearson's contingency chi-square test will be used to evaluate any differences between the randomization groups in opioid-related adverse events during the first 24-hour postoperative period.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Control - Fentanyl | Treatment - Methadone
Number analyzed (Participants) | 11 | 13
events
  Ondansetron Doses | 3.81 (1.70) | 3.43 (2.47)
  Emesis Episodes | 2.72 (2.45) | 2.08 (1.90)
  Hypoventilation Episodes | 0 (0) | 0 (0)
  Arrhythmias | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Control - Fentanyl | Treatment - Methadone
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control - Fentanyl (N=12) | Treatment - Methadone (N=14)
Postoperative Bleeding (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02747875/Prot_000.pdf